CLINICAL TRIAL: NCT02068144
Title: The Effect of Daily Dietary Supplementation With Cranberry Extract on Modulation of Cardiovascular Risk Factors in Obese, Insulin Resistant Human Subjects
Brief Title: The Effect of Cranberry Extract Supplementation on Cardiovascular Risk Factors in Obese, Insulin Resistant Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Ocean Spray, Inc. (Industry)
Responsible Party: Principal Investigator, Daniel Hsia, Principal and Medical Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PBRC 2013-047
Record Dates: First submitted 2014-02-18; First posted 2014-02-21 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Insulin Resistance; Atherosclerosis
Keywords: Cranberry Extract
MeSH Terms: conditions — Insulin Resistance; Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cranberry Extract (Experimental): Cranberry Extract in a 15.2oz beverage daily for 8 weeks
  Interventions: Dietary Supplement: Cranberry Extract
- Placebo (Placebo Comparator): Placebo 15.2oz beverage daily for 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Cranberry Extract — Participants will drink one 15.2 oz bottle of Cranberry Extract beverage daily for 8 weeks.
  Arms: Cranberry Extract
Other: Placebo — Participants will drink one 15.2oz bottle of placebo beverage daily for 8 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the health benefits of cranberry extract in people who are at risk for diabetes and heart problems.

DETAILED DESCRIPTION:
This study will be a double-blinded, randomized, placebo-controlled, pilot study in which subjects with pre-diabetes will be randomized to receive either placebo or Cranberry extract for a total of 8 weeks of treatment. Each subject will continue on the same dosage of cranberry extract or matching placebo for the entire duration of treatment. Comparisons for insulin sensitivity, endothelial function, and markers of inflmmation and oxidative stress will be made between the 2 groups pre and post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Are 20 years of age or older
* Not being treated with diabetes medication. However, if you are taking Metformin for pre-diabetes and are willing to stop taking the medication 2 weeks before and during the study that is ok. We will request clearance from your prescribing physician prior to stopping metformin and enrolling in the study.
* Have a blood sugar of 100-125 mg/dL (fasting) or 140-199 mg/dL after a 2 hour glucose tolerance test (determined by tests done at the screening visit)
* Have a fasting insulin more than or equal to 5 µIU/ml (determined by tests done at the screening visit)
* Have a Body Mass Index (BMI) ≥ 30 and ≤ 45.

Exclusion Criteria:

* Have a prior history of type 2 diabetes
* Are pregnant or breastfeeding.
* Are a woman able to have children and are not using birth control (i.e. barrier method, intrauterine and cervical devices, birth control pills, hormonal injections (Depo Provera® ), condoms with spermicidal gel or foam, contraceptive patch (Ortho Evra), diaphragm, or abstinence), or have had a tubal ligation or hysterectomy, or not at least 2 years past menopause.

  - All women able to have children will have a pregnancy test at the screening visit. If you become pregnant during the study, you will be dropped from the study.
* Have type 1 diabetes.
* Are taking steroids (except topical or inhaled steroids).

  - Other medications that may affect your blood sugar (i.e. certain blood pressure medications) are acceptable if the dose has not changed in the previous 6 months and the dose will not change during the study.
* Have a history or evidence of stomach or intestinal problems, e.g. irritable bowel syndrome; inflammatory bowel disease; ulcerative colitis or Crohn's disease; diverticulosis or diverticulitis; narrowing of the intestines, partial or complete removal of the stomach or small bowel; autonomic neuropathy consisting of difficulty swallowing; delayed stomach emptying or diarrhea; chronic, severe constipation; stomach or colon ulcers, or GI bleeding.
* Use laxatives or cathartics on a chronic basis.
* Take medications known to damage the kidneys, such as certain antibiotics, methicillin, and cyclosporin.
* Have any evidence of kidney disease.
* Have significant heart problems and/or history (within the last 6 months) of significant heart problems.
* Have evidence within the previous 6 months of liver disease such as hepatitis; jaundice; cirrhosis.
* Have clinically significant lung, neurologic, blood-related, immune system-related, cancer-related or metabolic disease.
* Have had a recurrence of cancer within the past five years, other than treated basal cell carcinoma.
* Are planning surgery during the study period.
* Have a history of substance abuse or alcoholism within the past 5 years, or significant psychiatric disorder that would interfere with your ability to complete the study.
* Have donated blood during the month before entering the study or are planning to donate blood during the study.
* Have participated in other studies using a research medication during the previous 3 months.
* Are currently smoking or have smoked within the past 6 months.

  - No smoking will be allowed during the study.
* Have had a fluctuation in body weight >5% in the previous 2 months.
* Are taking prescription or over-the-counter medication for weight loss.
* Are taking weight loss or herbal supplements.
* Are taking prescription or over-the-counter anti-inflammatory medications (such as naproxen, aspirin, ibuprofen).
* Are allergic to cranberries

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-02; Primary Completion 2016-06-02 (Actual); Study Completion 2018-07-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline Hyperinsulinemic-Euglycemic clamp at week 8 | 8 weeks +/- 2 days
  Insulin sensitivity is tested using a 120 mU/m2 hyperinsulinemic-euglycemic clamp at 100mg/dL glucose over 2 hours at weeks 0 and 8

SECONDARY OUTCOMES:
Change from baseline in endothelial function at week 7 | 8 weeks +/- 2 days
  Endothelial function by peripheral arterial tone (PAT) with an endo-PAT device prior to week 0 and week 7 as a surrogate measure of atherosclerosis.
Change from baseline in Indirect Calorimetry at week 8 | 8 weeks +/- 2 days
  Resting metabolic rate via indirect calorimetry will be measured using a Deltatrac II Metabolic cart at week 0 and week 8 as part of the hyperinsulinemic euglycemic clamp.
Change from screening to week 8 in lipid profile | 10 weeks +/- 2 days
  A comprehensive metabolic profile (CHEM 15) will be obtained at screening and then at week 8.
Change in body weight from baseline to week 8 | 8 weeks +/- 2 days
  Body weight will be assessed at baseline and week 8.
Change from screening to week 7 in oral glucose tolerance test (OGTT) | 8 weeks +/- 2 days
  A 2 hr OGTT will be performed prior to week 0 and at week 7
Change in nitric oxide level at baseline and week 8 | 8 weeks +/- 2 days
  Levels of nitric oxide will be assessed at baseline and after 8 weeks of intervention
Change in endothelin 1 level at baseline and week 8 | 8 weeks +/- 2 days
  Levels of endothelin 1 will be assessed at baseline and after 8 weeks of intervention
Change in oxidized LDL level at baseline and week 8 | 8 weeks +/- 2 days
  Levels of oxidized LDL will be assessed at baseline and after 8 weeks of intervention
Change in LOX-1 (Lectin-like oxidized low density lipoprotein-1) at baseline and week 8 | 8 weeks +/- 2 days
  Levels of LOX-1 (Lectin-like oxidized low density lipoprotein-1) will be assessed at baseline and after 8 weeks of intervention
Change in 8-isoprostanes at baseline and week 8 | 8 weeks +/- 2 days
  Levels of 8-isoprostanes will be assessed at baseline and after 8 weeks of intervention
Change in malondialdehyde at baseline and week 8 | 8 weeks +/- 2 days
  Levels of malondialdehyde will be assessed at baseline and after 8 weeks of intervention
Change in advanced glycation end products at baseline and week 8 | 8 weeks +/- 2 days
  Levels of advanced glycation end products will be assessed at baseline and after 8 weeks of intervention
Change in Apo A1 at baseline and week 8 | 8 weeks +/- 2 days
  Levels of Apo A1 will be assessed at baseline and after 8 weeks of intervention
Change in Paraoxonase at baseline and week 8 | 8 weeks +/- 2 days
  Levels of Paraoxonase will be assessed at baseline and after 8 weeks of intervention
Change in Adiponectin at baseline and week 8 | 8 weeks +/- 2 days
  Levels of Adiponectin will be assessed at baseline and after 8 weeks of intervention
Change in C-reactive protein (CRP) at baseline and week 8 | 8 weeks +/- 2 days
  Levels of C-reactive protein (CRP) will be assessed at baseline and after 8 weeks of intervention
Change in TNFα at baseline and week 8 | 8 weeks +/- 2 days
  Levels of TNFα will be assessed at baseline and after 8 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hsia, MD, Principal Investigator — Principal and Medical Investigator
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No